CLINICAL TRIAL: NCT05225324
Title: Equfina Tablet 50 mg Post Marketing Surveillance Protocol
Brief Title: A Post Marketing Surveillance Study of Equfina Tablet 50 Milligram (mg)
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: ME2125-M082-501
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Equfina
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Equfina 50 mg: Participants who will be prescribed with Equfina 50 mg tablets, orally within the scope of the approved label for Korea under the medical judgment of the investigator will be observed prospectively for 24 weeks.
  Interventions: Drug: Equfina 50 mg

INTERVENTIONS:
Drug: Equfina 50 mg — Equfina 50 mg tablets.

SUMMARY:
The purpose of this study is to describe the following in relation to the safety of Equfina Tablet 50 mg in the post marketing setting: 1. Serious adverse events (SAEs) and adverse drug reactions (ADRs) 2. Unexpected adverse events (AEs) and ADRs not reflected in the precautions for use 3. Known ADRs 4. Non-serious ADRs 5. Other safety and efficacy related information.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with idiopathic Parkinson's disease experiencing end of dose motor fluctuations who are receiving Equfina Tablet 50 mg as adjunctive treatment to levodopa-containing products
2. Participants who have given their consent to study participation about the use of personal data and medical data

Exclusion Criteria:

1. Participants taking over monoamine oxidase (MAO) inhibitors (example, selegiline hydrochloric acid [HCl], rasagiline mesylate)
2. Participants taking opioid drugs (example, pethidine HCl containing drugs, tramadol HCl containing products or tapentadol HCl)
3. Participants taking serotonergic drugs (example, tricyclic antidepressants, tetracyclic antidepressants, selective serotonin reuptake inhibitor, serotonin-noradrenaline reuptake inhibitors, selective noradrenaline reuptake inhibitor, noradrenergic and serotonergic antidepressant) or psychostimulant drugs (example, methylphenidate HCl, lisdexamfetamine dimesylate)
4. Participants taking dextromethorphan
5. Participants with severe hepatic impairment (Child-Pugh C)
6. Participants with a history of hypersensitivity to any of the ingredients of Equfina Tablet 50 mg
7. Pregnant women or women who may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants administered with Equfina Tablet 50 mg tablet will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With SAEs | From first dose of study drug up to 24 weeks
  A SAE is defined as any untoward medical occurrence: resulting in death; life threatening requiring hospitalization or prolongation of hospitalization; resulting in persistent or significant disability or incapacity; resulting in birth defect or congenital anomaly or medically important due to other reasons than above mentioned criteria.
Number of Participants With ADRs | From first dose of study drug up to 24 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Unexpected AEs | From first dose of study drug up to 24 weeks
  An AE is defined as any untoward and unintended signs (example, anomalies in laboratory test results) or symptoms/diseases occurring during administration/use of drugs, which do not necessarily have a causal relationship with the drug in question. An unexpected AE is an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug.
Number of Participants With Unexpected ADRs | From first dose of study drug up to 24 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs. An unexpected ADR is an ADR with difference in the nature or severity, specificity, or the outcome, compared to the product licensure/notification of the drug.
Number of Participants With Known ADRs | From first dose of study drug up to 24 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs. Known ADRs are those listed in product licensure/notification of the drug.
Number of Participants With Non-serious ADRs | From first dose of study drug up to 24 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.

SECONDARY OUTCOMES:
Change From Baseline in Score of Clinical Global Impression of Change (CGIC) | Baseline up to 24 weeks
  The CGIC is a 7-point scale that measures a physician's global impression of a participant's clinical condition. Scale ranges from 1 to 7 with lower scores indicating improvement (1=very much improved, 2=much improved, 3=minimally improved), higher scores indicating worsening (5=minimally worse, 6= much worse, 7=very much worse), and a score of 4 indicating no change.

CONTACTS AND LOCATIONS:
Locations (27):
- South Korea (27):
  - Site #23, Wŏnju, Gangwon-do
  - Site #11, Ilsan, Gyeonggi-do
  - Site #22, Yongin-si, Gyeonggi-do
  - Site #06, Cheonan, Gyeongsangnam-do
  - Site #09, Jinju, Gyeongsangnam-do
  - Site #07, Yangsan, Gyeongsangnam-do
  - Site #08, Iksan, Jeollabuk-do
  - Site #17, Jeonju, Jeollabuk-do
  - Site #18, Jeonju, Jeollabuk-do
  - Site #26, Jeonju, Jeollabuk-do
  - Site #03, Cheongju-si, North Chungcheong
  - Site #05, Busan
  - Site #16, Daegu
  - Site #25, Daegu
  - Site #20, Daejeon
  - Site #19, Gwanju
  - Site #24, Incheon
  - Site #02, Jeju City
  - Site #21, Sejong
  - Site #01, Seoul
  - Site #04, Seoul
  - Site #10, Seoul
  - Site #12, Seoul
  - Site #13, Seoul
  - Site #14, Seoul
  - Site #15, Seoul
  - Site #27, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.